CLINICAL TRIAL: NCT04153253
Title: Intravitreal Aflibercept Injection With Panretinal Photocoagulation Versus Early Vitrectomy for Diabetic Vitreous Hemorrhage
Brief Title: Intravitreal Aflibercept Injection or Early Vitrectomy for Diabetic Vitreous Hemorrhage
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Al Hadi Hospital (Other)
Responsible Party: Principal Investigator, Abeer MohamedSadeck Khattab, Abeer Mohamed Sadeck Khattab ,associate professor of ophthalmology., Al Hadi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 003-19
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Diabetic Vitreous Hemorrhage
Keywords: Aflibercept; panretinal photocoagulation; vitrectomy
MeSH Terms: interventions — aflibercept; Vitrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (Active Comparator): Intravitreal injection of Aflibercept followed by panretinal photocoagulation.
  Interventions: Drug: Aflibercept Injection [Eylea]
- Group II: Early vitrectomy. (Active Comparator): Early vitrectomy.
  Interventions: Procedure: Vitrectomy

INTERVENTIONS:
Drug: Aflibercept Injection [Eylea] — Three monthly based intravitreal injections were given followed by PRP if the hemorrhage was sufficiently cleared.Intravitreal injection was done in sterile operating room, after sterilization and toweling with application of sterile speculum, Betadine 5% drops was instilled into the conjunctiva and kept for two minutes followed by wash with balanced salt solution. Injection of 2mg /0.05m aflibercept was given 4 mm from the limbus in phakic eyes and 3.5 mm in pseudophakic with compression by sterile cotton tip on the site of injection, Paracentesis was done in cases of very high IOP following injection. At the end of procedure check of visual acuity was done (to be at least light perception).
  PRP was done if the hemorrhage is sufficiently cleared after the third injection.
  Arms: Group I
Procedure: Vitrectomy — Was done under local peribulbar anesthesia. After sterilization and toweling, wash with diluted betadine 5% was done. Insertion of three 23 valved cannulas beginning with the lower temporal one for infusion, clearance of anterior vitreous was done followed by core vitrectomy, peripheral vitrectomy , removal of posterior hyaloid aided by triamcinolone staining , trimming and removal of any vascular epicenters followed by vitreous base shaving with 360 scleral indentation, endolaser treatment was done for all eyes followed by fluid air exchange, 20% SF6 was used only if there is active significant bleeding during surgery or if there is intraoperative retinal tears, removal of cannulas was done at the end of surgery. All eyes received combination of topical steroid and antibiotic eye drops as postoperative treatment.
  Arms: Group II: Early vitrectomy.

SUMMARY:
Prospective study comparing efficacy and safety of intravitreal aflibercept injection and panretinal photocoagulation to early vitrectomy for patients with diabetic vitreous hemorrhage.

DETAILED DESCRIPTION:
Selected patients were divided into two groups, Group I for whom intravitreal aflibercept injection followed by panretinal photocoagulation was done and group II for whom early vitrectomy was done.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years.
* Any sex.
* Type Ι or ΙΙ DM,
* recent diabetic VH which is causing vision impairment, precluding complete PRP and needing treatment.
* BCVA is less than 20/70 (log MAR BCVA 0.6) and better than 20/1000 (log MAR BCVA 1.7).

Exclusion Criteria:

* Tractional retinal detachment.
* Previous PRP.
* History of anti VEGF therapy within the past two months.
* Neovascular glaucoma
* Subhyaloid hemorrhage.
* Vitreomacular traction.
* Diabetic macular edema .
* Patients with systemic contraindications for anti VEGF or unstable medical conditions as uncontrolled hypertension (persistently above 180/110 mmhg) or recent thromboembolic event within the past six months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-09-29 (Actual)

PRIMARY OUTCOMES:
Mean best corrected visual acuity(BCVA) change in both groups. | 9 months follow up.
  Final BCVA change measured in log MAR compared to initial BCVA.

SECONDARY OUTCOMES:
Rate of recurrent bleeding. | 9 months follow up.
  Rate of recurrent vitreous hemorrhage in both groups after initial clearance.
Number of additional treatment procedures . | 9 months follow up
  Additional treatment procedures done in cases of recurrent hemorrhage in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed H Abdelhamid, MD, Study Director — Alhadi hospital
Locations (1):
- Alhadi Hospital, Hawalli, Aljabyria, Kuwait

IPD SHARING:
Plan to Share IPD: Undecided
The data will be given from the author upon request.

REFERENCES:
- [Derived] Abd Elhamid AH, Mohamed AAEA, Khattab AM. Intravitreal Aflibercept injection with Panretinal photocoagulation versus early Vitrectomy for diabetic vitreous hemorrhage: randomized clinical trial. BMC Ophthalmol. 2020 Apr 6;20(1):130. doi: 10.1186/s12886-020-01401-4. PMID 32252674